CLINICAL TRIAL: NCT06879743
Title: Effect of Suboccipital Release on Neck Pain and Quality of Life in Patients With Fibromyalgia Syndrome
Brief Title: Effect of Suboccipital Release in Patients With Fibromyalgia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rowida Abd Elgleel Sayed Abd Elgleel, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Effect of suboccipital release
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected physiotherapy programme (Other)
  Interventions: Other: Suboccipital release
- Suboccipital release (Active Comparator)
  Interventions: Other: Suboccipital release

INTERVENTIONS:
Other: Suboccipital release — The ptients in this group recieve suboccipital release. The patient is positioned in a supine (lying on their back) position, allowing full relaxation of the cervical spine.
  The therapist places their fingertips or hands under the patient's occiput, making contact with the suboccipital muscles.
  Using gentle, sustained pressure, the therapist allows the weight of the head to create a release, often holding for 1-5 minutes.
  Subtle adjustments may be made, such as slight traction or rocking, to facilitate myofascial release and relaxation.

SUMMARY:
This study was designed to examine the efficacy of suboccipital release in Patients With FMS and to provide preliminary evidence regarding its effects on pain and QOL by objectively measuring Cortisol level in FMS patien

DETAILED DESCRIPTION:
Forty female patients with FM ( age : 20- 45 Years ) participated in the study after suing the consent form . Participants were randomly allocated assigned into 2 equal groups ( control group [ G1 ] and study [G2 ] ) . Group

1 received selected physical therapy programme. Group 2 recieved suboccipital release. All participants were assessed for cortisol and pain level by using visual analogues scale and neck disability scale. Also participants were assessed by pressure algometer for pain intensity. Participants were assessed for QOL by FIBROMYALGIA IMPACT QUESTIONNAIRE (FIQR) . treatment was done 3 sessions per weeks for successive 6 weeks pre and post assessment for all valuable were Done

ELIGIBILITY:
Inclusion Criteria:

* women between 20-45 years old, (ii) diagnoses according to the 2016

American College of Rheumatology criteria for fibromyalgia [1]

* Symptoms have been present at a similar level for at least three months (iii) Absence of other disorders that causes similar symptoms: systemic lupus erethromatosis (SLE), rheumatoid arthritis (RA) and Lyme disease based on laboratory investigations (erythrocyte sedimentation rate (ESR), Anti anti-cyclic citrullinated peptide (Anti CCP), antinuclear antibody (ANA) and Rheumatoid factor(RF)).
* Exclusion Criteria:

  * any medical, neurological, or psychiatric illness, use of strong opioids or other painkillers except paracetamol and/or ibuprofen, benzodiazepine, illicit drug or alcohol use, recent use of cannabis, pregnancy, breast feeding, and the presence of pain syndromes other than FM. Presence of other autoimmune disorders e.g.: rheumatoid arthritis and systemic lupus erethromatosus

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Cortisol level | Six weeks after begining of intervention
  Changes in pain from baseline to six weeks after begining of intervention

SECONDARY OUTCOMES:
Fibromyalgia impact questionair | Six weeks after begining of intervention
  Changes of quality of life from baseline to six weeks after begining of interventio

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy laps at cairo university, Cairo, Egypt